CLINICAL TRIAL: NCT05510622
Title: Reproductive Tract Microbiome in Women With Recurrent Pregnancy Loss
Brief Title: Uterine Microbiome in Recurrent Pregnancy Loss
Status: Recruiting | Type: Observational
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 05/22/DD-BVMD
Record Dates: First submitted 2022-08-13; First posted 2022-08-22 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Pregnancy Loss, Not Pregnant; Vaginal Microbiome
Keywords: Microbiome; Recurrent Pregnancy Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Microbiome analysis using 16S ribosomal RNA sequencing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Recurrent pregnancy loss: Women with history of recurrent pregnancy loss
  Interventions: Other: Vaginal swab and endometrial biopsy
- Control: Normal fertile women
  Interventions: Other: Vaginal swab and endometrial biopsy

INTERVENTIONS:
Other: Vaginal swab and endometrial biopsy — A vaginal swab (DNA/RNA shield collection tube with swab - Zymo Research, CatNo R1107) and endometrial biopsy (Endobrush® - Lab CCD, Paris, France) will be obtained during 18th - 22nd day of the menstrual cycle.

SUMMARY:
The female genital tract microbiome may reflect female reproductive health and may be related to pregnancy outcomes. Disturbances in this microbiome may be associated with adverse reproductive outcomes. The investigators hypothesize that the endometrial and vaginal microbiome composition in women with a history of recurrent pregnancy loss are different, compared with those in normal fertile women.

DETAILED DESCRIPTION:
The investigators want to describe the endometrial microbiome composition in normal fertile women and women with a history of recurrent pregnancy loss by analyzing mid-luteal phase vaginal swab and endometrial biopsy samples using 16S rRNA sequencing.

ELIGIBILITY:
1. Recurrent pregnancy loss patients

   Inclusion Criteria:
   * 18-38 years old
   * Having a regular menstrual cycle, from 25 to 35 days
   * Having ≥ 2 recurrent pregnancy loss and
   * Couples with normal karyotype results
   * Having no condition causing pregnancy loss such as antiphospholipid syndrome, abnormal thyroid function.
   * Agree to participate in the study

   Exclusion Criteria:
   * Irregular menstrual cycle
   * Having uterine abnormalities (e.g., adenomyosis, intrauterine adhesions, unicornuate/ bicornuate/ arcuate uterus; unremoved hydrosalpinx, endometrial polyp, submucosal fibroid)
   * Using intrauterine device within the last 3 months
   * Using antibiotic/vaginal pessary/contraceptive pills within 2 weeks
   * Having sexual intercourse within 48 hours
2. Healthy control patients

Inclusion Criteria:

* 18-38 years old
* Having a regular menstrual cycle, from 25 to 35 days
* No history of pregnancy loss
* Having 1 or more live birth, with the youngest child ≥ 6 months old
* Agree to participate in the study

Exclusion Criteria:

* Irregular menstrual cycle
* Having uterine abnormalities (e.g., adenomyosis, intrauterine adhesions, unicornuate/ bicornuate/ arcuate uterus; unremoved hydrosalpinx, endometrial polyp, submucosal fibroid)
* Using intrauterine device within the last 3 months
* Using antibiotic/vaginal pessary/contraceptive pills within 2 weeks
* Having sexual intercourse within 48 hours

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: For RPL women: having ≥ 2 recurrent pregnancy loss. For NF women: having ≥ 1 live birth, with no history of pregnancy loss
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Midluteal bacterial composition of endometrium in women with recurrent pregnancy loss and control group | 1 week
  Bacterial composition in the endometrium in midluteal phase are analysed using 16S rRNA gene sequencing

SECONDARY OUTCOMES:
Midluteal bacterial composition of vagina in women with recurrent pregnancy loss and control group | 1 week
  Bacterial composition in the vaginal in midluteal phase are analysed using 16S rRNA gene sequencing
Phylogenetic tree of endometrial microorganisms in women with recurrent pregnancy loss and control group | 1 week
  Phylogenetic tree based on 16S rRNA gene sequences
Phylogenetic tree of vaginal microorganisms in women with recurrent pregnancy loss and control group | 1 week
  Phylogenetic tree based on 16S rRNA gene sequences

CONTACTS AND LOCATIONS:
Overall Officials: Lan N Vuong, MD, PhD, Study Chair — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (2):
- Vietnam (2):
  - My Duc Hospital, Ho Chi Minh City, Ho Chi Minh City
  - My Duc Phu Nhuan Hospital, Ho Chi Minh City, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Undecided